CLINICAL TRIAL: NCT04049045
Title: Effects of Empagliflozin on Diuresis and Renal Function in Patients With Acute Decompensated Heart Failure
Acronym: EMPAG-HF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Christian Schulze (Other)
Collaborators: Boehringer Ingelheim (Industry); Zentrum für Klinische Studien Jena (Other)
Responsible Party: Sponsor-Investigator, Christian Schulze, Prof. Dr. med. P. Christian Schulze, Jena University Hospital
Organization: Jena University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZKSJ0109
Record Dates: First submitted 2019-07-10; First posted 2019-08-07 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Acute Decompensated Heart Failure
Keywords: acute decompensated heart failure; empagliflozin; diuresis; renal function
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, double-blind, placebo-controlled, randomized and interventional exploratory study
Who Masked: Participant, Care Provider, Investigator
Masking Description: There will be two trial medications, the licensed medicinal product empagliflozin, trade name Jardiance®, 25 mg and matching placebo tablets. The placebo tablets will be indistinguishable by appearance, taste, smell, weight from the investigational product. Both will be stored in plastic containers containing 30 tablets each.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum arm (Active Comparator): 25 mg tablet of empagliflozin once daily for five days
  Interventions: Drug: Empagliflozin 25 mg
- Placebo arm (Placebo Comparator): one tablet of the matching Placebo once daily for five days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 25 mg — Empagliflozin 25 mg film-coated tablets, for oral use administered once daily for 5 days in addition to routinely administered (weight adjusted) intravenous furosemide
  Arms: Verum arm
Drug: Placebo — matching Placebo, film-coated tablets, for oral use, matching to investigational product Jardiance® administered once daily for 5 days in addition to routinely administered (weight adjusted) intravenous furosemide
  Arms: Placebo arm

SUMMARY:
Heart failure is the most common hospital admission diagnosis and shows increasing incidence and prevalence in Germany, the United States and worldwide. Improvements in the primary treatment conditions for e.g. myocardial infarction and reduced primary mortality has resulted in an increasing group of patients with secondary cardiac abnormalities including chronic heart failure.

Progressive cardiac dysfunction and failure are associated with exercise intolerance, volume retention, nocturia, dyspnoea among others. The most severe progression of heart failure is cardiac decompensation (also called: acute heart failure) and cardiogenic shock. Volume retention, abnormal renal function and diuretic resistance are hallmarks of this clinical phenotype. Currently, the only available treatment is diuresis through various combinations of diuretics and the addition of cardiac inotropes when cardiac hypoperfusion is documented. Patients with acute decompensated heart failure (ADHF) often develop a state of diuretic resistance characterized by a need of rising dosages of diuretics for adequate diuresis and urine production.

ADHF patients also show metabolic abnormalities including insulin resistance or type 2 diabetes mellitus.

Empagliflozin is a potent and selective inhibitor of the sodium glucose cotransporter 2 (SGLT2) used in the treatment of type 2 diabetes. By inhibiting SGLT2, empagliflozin reduces renal glucose reabsorption and increases urinary glucose excretion. In addition to reducing hyperglycaemia, empagliflozin is associated with osmotic diuresis, reductions in weight and blood pressure without increases in heart rate, and has favourable effects on markers of arterial stiffness and vascular resistance.

The investigators propose a single center exploratory study to test the hypothesis that the application of empagliflozin in addition to standard diuretic regimens increases urine output, decreases the need for further acceleration of diuretic regimens, and positively influences renal function as well as metabolism including insulin resistance in ADHF patients. Thereby, empagliflozin may be effective in the prevention of complex cardio metabolic alterations involved in ADHF.

DETAILED DESCRIPTION:
If feasible (run-in of patients into the hospital from 08:00 a.m. to 06:00 p.m.) screening/baseline, enrolment, randomization and first dose of empagliflozin should be performed on the same day. In general, but especially in case of other run-in times (e.g. late evening, night and early morning hours) screening/baseline time period should not exceed 12 hours. In case a patient has to spend the night in hospital before randomization can be executed, a time period of up to 16 hours will not be counted as protocol deviation.

ELIGIBILITY:
Inclusion Criteria:

* Patients (age between 18-85 years) with acute decompensated heart failure (HF).
* Brain Natriuretic Peptide (BNP) >100 pg/ml, or N-terminal pro-BNP (NT-proBNP)>300 pg/ml as defined by current clinical guidelines for the diagnosis of acute decompensated HF (European Society of Cardiology 2016 HF guideline)
* Patients with diabetes mellitus type 2 or impaired glucose tolerance as defined by current clinical guidelines (German and International Diabetes Society 2016: HbA1c>6.5 % (upper limit for this clinical trial 12 %) or fasting glucose >7.0 mmol/l or any incidental glucose level >11.1 mmol/l or abnormal oral glucose tolerance test with 2h plasma glucose >7.8 mmol/l) or on antidiabetic medication or antidiabetic diet or patients with normal Glucose tolerance
* Patients without cognitive impairment, i.e. they must be capable of understanding the nature, significance and implications of the clinical trial and to form a rational intention in the light of the facts
* Written informed consent obtained
* For women with childbearing potential (until 2 years after menopause):

  * Negative pregnancy test
  * regular and correct use of a highly effective contraceptive method with an error rate of <1% per year (e.g. combined (estrogen and progesteron) hormonal contraception (oral, intravaginal, transdermal), progesteron-only hormonal contraception (oral, injectable, implantable), intrauterine device (IUD), intrauterine hormone-releasing system (IUS) tubal ligation (female sterilization), hormon donating intrauterine device ("hormonal spiral"), double barrier methods, sexual abstinence, vasectomy of the partner)

Exclusion Criteria:

* Type 1 diabetes mellitus
* Chronic Kidney Disease (CKD) with eGFR< 30 ml/min, or end-stage renal failure with the need for chronic dialysis treatment
* Acute kidney injury (AKI) ≥ Acute Kidney Injury Network (AKIN) stage 2 or requiring dialysis treatment
* Current medication with SGLT-2 inhibitors
* Known intolerance or hypersensitivity to the active substance empagliflozin, lactose or any other of the excipients listed in section 6.1. of the summary of product characteristics (SmPC). A contraindication or intolerance to furosemide
* Acute heart failure without signs of congestion ("dry" patient)
* Indication for urgent coronary angiography or any planned administration of a iodine based contrast agent within the next 6 days
* Need for hemofiltration or any other form of extracorporeal therapy
* Planned surgery
* Previous participation in this trial or recent participation in another clinical trial (within the last 3 months before inclusion, so that medical product/s from previous trial participation/s have been fully washed out )Identification of any causes of heart failure leading to decompensation that needs urgent management (like acute coronary syndrome, severe unstable arrhythmias, mechanical causes, acute pulmonary embolism)
* Incapacity to understand and / or to provide written informed consent
* Ongoing reported alcohol abuse (daily alcohol intake of more than 2 drinks (liquor, beer or wine) in men and 1 drink in women, corresponding to 12/24 g of pure alcohol per day women / men and/ or obvious alcoholisation of the patient during screening )

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-29 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Total urinary output (UOP) as measured by daily volume summed up over 5 days | 5 days
  Total UOP as summed over 5 days

SECONDARY OUTCOMES:
Renal function under treatment | 5 days
  Change of creatinine values: increase in creatinine of > 0.3 mg/dl, doubling of serum creatinine, need for renal replacement therapy
Net fluid output | 5 days
  UOP - fluid intake
Worsening or persistent heart failure | 30 days
  NYHA class (New York Heart Association functional heart failure classification)
Intermediate Care (IMC) / Intensive Care Unit (ICU) and hospital length of stay | 30 days
  Duration in days
Liver function | 30 days
  bilirubin, serum aminotransferases, relevant change in coagulation status
Pulmonary function | 30 days
  oxygen saturation without oxygen therapy/ need for oxygen in l/min, presence of rales, changes in chest x-ray (worsening/ improvement/ new infiltration)
Number of patients alive and out of hospital -after 30 days | 30 days
  number of patients

OTHER OUTCOMES:
Safety Outcome: Number of Adverse Events and Serious Adverse Events including MedDRA-SAE Preferred Terms and SOCs in both groups | 30 days
  Listing of all adverse events and serious adverse events, laboratory parameters as far as not efficacy parameters

CONTACTS AND LOCATIONS:
Overall Officials: Christian Schulze, Prof. Dr., Principal Investigator — Department of Internal Medicine I, Jena University Hospital
Locations (1):
- Department of Internal Medicine I, Jena University Hospital, Jena, Germany

REFERENCES:
- [Derived] Schulze PC, Bogoviku J, Westphal J, Aftanski P, Haertel F, Grund S, von Haehling S, Schumacher U, Mobius-Winkler S, Busch M. Effects of Early Empagliflozin Initiation on Diuresis and Kidney Function in Patients With Acute Decompensated Heart Failure (EMPAG-HF). Circulation. 2022 Jul 26;146(4):289-298. doi: 10.1161/CIRCULATIONAHA.122.059038. Epub 2022 Jun 29. PMID 35766022